CLINICAL TRIAL: NCT00363428
Title: A Randomized Trial of Pulmonary Rehabilitation in Patients With Moderate to Severe COPD Who Require Lung Resection for Lung Cancer
Brief Title: Lung Rehabilitation in Treating Patients With Chronic Obstructive Pulmonary Disease Who Are Undergoing Surgery for Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MC0825; P30CA047904 (NIH); K23CA106544 (NIH); 08-007135 (Other: Mayo Clinic IRB); NCI-2009-01148 (Registry Identifier: NCI-CTRP); MC0825 (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Lung Cancer; Perioperative/Postoperative Complications; Pulmonary Complications; Tobacco Use Disorder
Keywords: pulmonary complications; perioperative/postoperative complications; tobacco use disorder; non-small cell lung cancer; small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Postoperative Complications; Tobacco Use Disorder; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Counseling; Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Receive standard care and educational material on exercise and lifestyle choices of well-being
  Interventions: Behavioral: exercise intervention; Behavioral: smoking cessation intervention; Other: counseling intervention; Other: educational intervention; Procedure: conventional surgery; Procedure: pulmonary complications management/prevention
- Lifestyle intervention (Experimental)
  Interventions: Behavioral: exercise intervention; Behavioral: smoking cessation intervention; Other: counseling intervention; Other: educational intervention; Procedure: conventional surgery; Procedure: pulmonary complications management/prevention

INTERVENTIONS:
Behavioral: exercise intervention — life style
Behavioral: smoking cessation intervention — Life style
Other: counseling intervention — life style
Other: educational intervention — life style
Procedure: conventional surgery — life style
Procedure: pulmonary complications management/prevention — life style

SUMMARY:
RATIONALE: Exercise may help improve lung function and lessen complications of surgery in patients with chronic obstructive pulmonary disease who are undergoing surgery for lung cancer. It is not yet known whether lung rehabilitation is more effective than standard therapy in improving lung function in patients with chronic obstructive pulmonary disease who are undergoing surgery for lung cancer.

PURPOSE: This randomized clinical trial is studying lung rehabilitation to see how well it works compared to standard therapy in treating patients with chronic obstructive pulmonary disease who are undergoing surgery for lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the impact of preoperative pulmonary rehabilitation (including upper and lower extremity resistance training) vs usual care in patients with lung cancer and moderate to severe chronic obstructive pulmonary disease who require lung resection for lung cancer.
* Compare the impact of this study intervention vs usual care on functional status after surgery.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 intervention arms.

* Arm I: Patients undergo pulmonary rehabilitation (including daily upper and lower extremity resistance training, education, and smoking cessation counseling) twice a day for 5 days prior to surgical resection. Beginning 2-3days after surgery, patients undergo pulmonary rehabilitation once a day until discharge from the hospital.
* Arm II: Patients receive usual care (education and smoking cessation counseling alone) twice a day for 5 days prior to surgical resection. Following surgery, patients will receive usual care once a day until discharge from the hospital.

Days of hospitalization, ICU admissions, postoperative complications (i.e., pneumonia, mechanical ventilation > 48 hours, or atelectasis requiring bronchoscopy) and spirometry and imaging studies will be evaluated after surgery.

After completion of study intervention, patients are followed at 4-6 weeks, at 12 weeks, and at 6 months.

PROJECTED ACCRUAL: A total of 90 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of lung cancer
* Scheduled to undergo any thoracotomy for lung cancer resection (including wedge) or VATS lobectomy or pneumonectomy for lung resection
* Diagnosis of COPD, meeting the following criteria:

  * FEV_1/FVC < 0.71
  * Smoking history ≥ 10 pack/years
* Presence of moderate to severe lung disease, meeting 1 of the following:

  * FEV_1 ≤ 60% predicted*
  * FEV_1< 80% predicted AND significant shortness of breath defined by a score of 2 or higher in the Medical Research Council Dyspnea Score NOTE: *Patients with an FEV1 < 60% predicted (most severe) and scheduled to undergo VATS segmentectomy or wedge resection will also be included.

PATIENT CHARACTERISTICS:

* Able to physically utilize exercise equipment as part of rehabilitation program
* No poor motivation or likely not to participate fully in PR program
* No recent history (within the past 3 months) of a clinically-significant myocardial infarction, unstable angina, serious cardiac arrhythmia, or other serious medical condition which the attending physician performing the preoperative evaluation deems incompatible with participation in the study

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 40 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2012-11-01 (Actual); Study Completion 2012-11-01 (Actual)

PRIMARY OUTCOMES:
Length of stay in hospital and functional status measured at 12 weeks post-operatively | 12 weeks

SECONDARY OUTCOMES:
Hospital re-admission | 12 months
Oxygen requirement | 12 months
Post-operative pulmonary function | 12 months
Respiratory care interventions | 12 months
Number and percentage of patients with postoperative complications (defined as pneumonia, mechanical ventilation of more than 2 days, or atelectasis requiring a bronchoscopy) | 12 months
Measured physical activity at 6 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto P. Benzo, MD, MS, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Perrotta F, Cennamo A, Cerqua FS, Stefanelli F, Bianco A, Musella S, Rispoli M, Salvi R, Meoli I. Effects of a high-intensity pulmonary rehabilitation program on the minute ventilation/carbon dioxide output slope during exercise in a cohort of patients with COPD undergoing lung resection for non-small cell lung cancer. J Bras Pneumol. 2019 Oct 14;45(6):e20180132. doi: 10.1590/1806-3713/e20180132. eCollection 2019. PMID 31618297